CLINICAL TRIAL: NCT03055325
Title: Post-surgery Systemic Inflammation and Neuro-immune Interactions
Acronym: POSINI
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lars I Eriksson, Professor, Senior Consultant, Karolinska University Hospital
Other Study IDs: POSINI
Record Dates: First submitted 2017-01-10; First posted 2017-02-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Inflammation; Surgery
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical patients: Cognitive testing, testing of heart rate variability and collection of blood samples
  Interventions: Other: Observational study of patients undergoing surgery

INTERVENTIONS:
Other: Observational study of patients undergoing surgery — Cognitive testing, testing of heart rate variability and collection of blood samples

SUMMARY:
The aim is to map the inflammatory response after surgery and further investigate the mechanisms by which inflammation is regulated. The inflammatory cascade is pivotal in protecting organisms against invading pathogens and in enabling healing of damaged tissues, yet the cascade itself may be harmful to the organism when excessive (e g septic chock).

The increased immune-reactivity after trauma, such as surgery, is furthermore associated with post-operative declines in memory and learning capacity, a condition likely related to the notion of "sickness behavior". The effects on the brain after surgery and the associated neuro-immune crosstalk will now be investigated with focus on changes in immune reactivity in peripheral blood after surgery.

DETAILED DESCRIPTION:
Surgical trauma causes release of damage-associated molecular patterns (DAMPs) and other alarmines (e.g. high mobility group box (HMGB-1)) targeting receptors on local cells of the innate immune system, such as macrophages. This cellular response to trauma is followed by a rapid release of an array of inflammatory mediators (e.g. tumor necrosis factor alfa (TNFa), interleukin (IL)-1B, IL-6, IL-8, IL-10) being dependent on intracellular activation of nuclear factor nuclear factor kappa beta (NF-kB). Until recently it was believed that the brain is protected from this cascade of inflammatory mediators primarily due to an intact blood-brain-barrier (BBB). However, there is now a growing body of evidence that long term impairment of brain functions is associated with trauma-induced activation of the brain innate immune system with subsequent impairment of higher cognitive processes and risk for later permanent dementia. Yet, the link between systemic inflammation and cognitive impairment is not fully understood.

A recent study has mapped periphery-to-brain-signaling after surgical trauma and the impact of major surgical trauma on the human brain by serial positron emission tomography (PET)-imaging. In series of surgical patients, profound and biphasic changes in brain immune activity after surgery has been demonstrated after major abdominal surgery with signs of early depression followed by an increased immune activity at 3 months postoperatively. These biphasic changes in brain immunity seem to be aligned with simultaneous changes in whole blood immune reactivity to lipid polysaccharide (LPS) suggesting a close link between brain and peripheral immune systems in regulation of acute inflammation and immune responses. Preclinical work in surgical animal models indicates disruption of the BBB with migration of peripheral macrophages into the brain as a pathway of potential importance. Evidence from an orthopedic surgery model in mice of trauma-induced altered hippocampal neuro-immune activity further raises the question whether peripheral markers of neurodegeneration S100b, neurofilament light (NFL), ptau, beta-amyloid) are associated with postoperative cognitive dysfunction (POCD).

The immune-regulatory role of the brain via the cholinergic anti-inflammatory reflex pathway (mediated by the vagal nerve) has been identified as potential target for immune-modulatory treatment strategies in systemic inflammation. We have moreover demonstrated a distinct release of human carotid body inflammatory mediators at hypoxia and gene expression related to inflammatory mediators, suggesting a potential role of the human carotid body in periphery-to-brain immune-signaling. Modulation of a vagal nerve-derived inflammatory reflex pathway by electrical stimulation has recently been successfully applied in treatment of chronic inflammation among patients with rheumatoid arthritis.

The hypothesis is that vagal nerve activity modulates systemic inflammation in patients after major surgery and that this modulation is associated with cognitive performance in the postoperative period.

With a more comprehensive understanding of immune-to-brain signaling after surgical trauma and how this biphasic inflammatory response pattern is regulated by cellular and neuronal components, the impact of immune modulation on key processes behind surgery-induced brain dysfunction can be explored, and possible neural and humoral targets for relevant anti-inflammatory treatments established.

ELIGIBILITY:
Inclusion Criteria:

* Male
* BMI <33
* Age 45-75
* No significant neurological, cardiovascular or rheumatic diseases
* Mini-mental state examination (MMSE) >23

Exclusion Criteria:

* Unable to understand informed concent
* Medication with Statins, beta blockers or immunomodulatory drugs

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective abdominal surgery
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
TNF alpha in blood | After LPS provocation within 4 hours
  Ex vivo

SECONDARY OUTCOMES:
Immune cells and inflammatory markers in peripheral blood | Before surgery and up to 12 months after surgery
Heart rate variability | Before surgery and up to 6 months after surgery
Cognitive testing using the International Study of Post-Operative Cognitive Dysfunction | Before surgery and up to 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lars I Eriksson, Principal Investigator — Department of Physiology and Pharmacology, Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided